CLINICAL TRIAL: NCT07027709
Title: Clinical Performance of Hybrid Ceramic Laminate Veneers With Two Pretreatment Protocols: A Randomized Clinical Trial
Brief Title: Clinical Performance of Hybrid Ceramic Laminate Veneers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Omnia Mohammed Wafik, PRINCIPLE INVESTIGATOR, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CU-FP-HCLV-001
Record Dates: First submitted 2025-06-11; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Bonding of Veneers After Different Treatment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BeautiBond Xtreme Pretreatment Group (Experimental): atients in this group will receive laminate veneers fabricated from HC hard blocks. The inner surface of the veneers will be pretreated with BeautiBond Xtreme, and the veneers will be bonded using BeautiLink SA self-adhesive resin cement. This group is used to assess the clinical performance of BeautiBond Xtreme pretreatment over an 18-month follow-up.
  Interventions: Device: BeautiBond Xtreme pretreatment with BeautiLink SA cementation
- HC Primer Pretreatment Group (Active Comparator): atients in this group will receive laminate veneers fabricated from HC hard blocks. The inner surface of the veneers will be pretreated with HC Primer, and the veneers will be bonded using BeautiLink SA self-adhesive resin cement. This group serves as a comparator to evaluate differences in clinical outcomes relative to the BeautiBond Xtreme group.
  Interventions: Procedure: HC Primer pretreatment with BeautiLink SA cementation

INTERVENTIONS:
Device: BeautiBond Xtreme pretreatment with BeautiLink SA cementation — Laminate veneers fabricated from HC hard blocks were pretreated on the internal surface with BeautiBond Xtreme, then bonded to tooth structure using BeautiLink SA self-adhesive resin cement. The tooth surfaces were also treated with BeautiBond Xtreme. Veneers were digitally designed and milled, then cemented following a standardized clinical protocol.
  Arms: BeautiBond Xtreme Pretreatment Group
Procedure: HC Primer pretreatment with BeautiLink SA cementation — Laminate veneers fabricated from HC hard blocks were pretreated on the internal surface with HC Primer, then bonded to tooth structure using BeautiLink SA self-adhesive resin cement. The tooth surfaces were treated with BeautiBond Xtreme. Veneers were digitally designed and milled, then cemented following the same clinical protocol used in the experimental grou
  Arms: HC Primer Pretreatment Group

SUMMARY:
This randomized controlled trial evaluates the clinical performance of laminate veneers fabricated from HC hard blocks pretreated with BeautiBond Xtreme versus HC Primer, using BeautiLink SA cement. The study focuses on marginal adaptation, retention, discoloration, and recurrent caries over 18 months.

DETAILED DESCRIPTION:
This clinical trial compares two bonding protocols for hybrid ceramic laminate veneers. The veneers are fabricated from HC hard blocks and bonded using BeautiLink SA resin cement. One group receives BeautiBond Xtreme pretreatment, while the other receives HC Primer. The study assesses marginal adaptation, retention, recurrent caries, and discoloration over 18 months to determine the superior clinical bonding protocol for these restorations.

ELIGIBILITY:
Inclusion Criteria:dult patients ≥ 21 years requiring laminate veneers in the esthetic zone, vital or endodontically treated teeth, sufficient enamel, willing and able to consent and comply.

-

Exclusion Criteria: Periodontal disease, bruxism, poor hygiene, pregnancy, systemic illness, allergies, insufficient enamel, ongoing trials, orthodontic treatment.

-

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome: Marginal Adaptation | Measured at 6, 12, 18 months.
  (Modified USPHS)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
this is a university-sponsored clinical study with a small sample size and limited scope. No plan to share individual participant data (IPD) has been established due to privacy considerations and the nature of the trial. However, summary-level results may be published in peer-reviewed journals and conferences.

REFERENCES:
- [Result] Çötert İ, Çötert HS. Survival of partial laminate veneers and categorical covariates affecting the survival: a systematic review. Open Dent J. 2023;17(1) Ho CCK. Appraisal and cementation of porcelain laminate veneers. In: Banerji S, Mehta SB, Ho CCK, editors. Practical procedures in aesthetic dentistry. West Sussex: John Wiley & Sons; 2017. Bajaj M, Jha P, Nikhil V. Shade selection in esthetic dentistry. IP Indian J Conserv Endod. 2023;8(2):79-85. http://doi. org/10.18231/j.ijce.2023.015. De Munck, J., Van Landuyt, K., Peumans, M., Poitevin, A., Lambrechts, P., Braem, M., & Van Meerbeek, B. (2012). A critical review of the durability of adhesion to tooth tissue: methods and results. Journal of Dental Research, 91(4), 351-381. Frankenberger, R., Hartmann, V. E., Krech, M., Krämer, N., Reich, S., Braun, A., & Roggendorf, M. (2015). Adhesive luting of new CAD/CAM materials. International Journal of Computerized Dentistry, 18(1), 9-20. Morimoto, S., Rebello de Sampaio, F. B., Braga, M. M., Sesma, N., & Özcan, M. (2016). Survival rate of resin and ceramic inlays, onlays, and overlays: a systematic review and meta-analysis. Journal of Dental Research, 95(9), 985-994. Lawson, N. C., Bansal, R., & Burgess, J. O. (2016). Wear, strength, modulus and hardness of CAD/CAM restorative materials. Dental Materials, 32(11), e275-e283. El Zohairy, A.A.; De Gee, A.J.; Mohsen, M.M.; Feilzer, A.J. Microtensile bond strength testing of luting cements to prefabricated CAD/CAM ceramic and composite blocks. Dent. Mater. 2003, 19, 575-583.Lührs, A. K., De Munck, J., Geurtsen, W., & Van Meerbeek, B. (2014). Composite cements benefit from light-curing. Dental Materials, 30(3), 292-301. Frankenberger, R.; Lohbauer, U.; Taschner, M.; Petschelt, A.; Nikolaenko, S.A. Adhesive luting revisited: influence of adhesive, temporary cement, cavity cleaning, and curing mode on internal dentin bond strength. J. Adhes. Dent. 2007, 9, 269-273. Dos Santos, V.H.; Griza, S.; de Morae